CLINICAL TRIAL: NCT02520739
Title: New Industrial Procedures for Achieving a Nutritional Added Value of the Olive Oil. The NUTRAOLEUM Study
Acronym: NUTRAOLEUM
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fundación Pública Andaluza para la Investigación Biomédica Andalucía Oriental (Other)
Collaborators: Hospital del Mar (Other); Instituto de Nutrición y Tecnología de los Alimentos (Other)
Responsible Party: Principal Investigator, Sarah Biel, HEAD OF PROJECT MANAGEMENT, Fundación Pública Andaluza para la Investigación Biomédica Andalucía Oriental
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 13/11-C38
Record Dates: First submitted 2014-11-28; First posted 2015-08-13 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-03

CONDITIONS: Cardiovascular Diseases
Keywords: olive oil; phenolic compounds; triterpenes; oxidation and inflammation
MeSH Terms: conditions — Cardiovascular Diseases; Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Virgin Olive Oil (Placebo Comparator): Virgin olive oil obtained by traditional procedures (VOO);
  Interventions: Dietary Supplement: Virgin Olive Oil (VOO)
- Optimized High Phenolic Content Oil (Experimental): Optimized virgin olive oil with a high phenolic content (OHPCO);
  Interventions: Dietary Supplement: Optimized High Phenolic Content Oil (OHPCO)
- Functional Olive Oil (Experimental): Functional olive oil (FOO) with both high phenolic compounds and triterpene content.
  Interventions: Dietary Supplement: Functional Olive Oil (FOO)

INTERVENTIONS:
Dietary Supplement: Virgin Olive Oil (VOO) — VOO was sequentially administered over 3 periods of 3 weeks preceded by 2-week washout periods in which participants were requested to avoid olives and olive oil consumption. During intervention periods, they were requested to ingest a raw daily dose of 30 mL of VOO distributed over 3 meals. Daily doses of VOO were blindly prepared in special containers, with the corresponding 30 mL VOO daily dose were delivered at the beginning of each intervention period to the participants. The participants were instructed to return the containers when collecting the next daily doses for the amount of unconsumed VOO to be registered. During washout periods participants were provided of sunflower oil for raw and cooking purposes.
  Arms: Virgin Olive Oil
Dietary Supplement: Optimized High Phenolic Content Oil (OHPCO) — OHPCO was sequentially administered over 3 periods of 3 weeks preceded by 2-week washout periods in which participants were requested to avoid olives and olive oil consumption. During intervention periods, they were requested to ingest a raw daily dose of 30 mL of OHPCO distributed over 3 meals. Daily doses of OHPCO were blindly prepared in special containers, with the corresponding 30 mL OHPCO daily dose were delivered at the beginning of each intervention period to the participants. The participants were instructed to return the containers when collecting the next daily doses for the amount of unconsumed OHPCO to be registered. During washout periods participants were provided of sunflower oil for raw and cooking purposes.
  Arms: Optimized High Phenolic Content Oil
Dietary Supplement: Functional Olive Oil (FOO) — FOO was sequentially administered over 3 periods of 3 weeks preceded by 2-week washout periods in which participants were requested to avoid olives and olive oil consumption. During intervention periods, they were requested to ingest a raw daily dose of 30 mL of FOO distributed over 3 meals. Daily doses of FOO were blindly prepared in special containers, with the corresponding 30 mL FOO daily dose were delivered at the beginning of each intervention period to the participants. The participants were instructed to return the containers when collecting the next daily doses for the amount of unconsumed FOO to be registered. During washout periods participants were provided of sunflower oil for raw and cooking purposes.
  Arms: Functional Olive Oil

SUMMARY:
The Mediterranean diet, in which olive oil is the main source of fat, has shown to be protective for chronic degenerative diseases. These diseases, such as cardiovascular, cancer, and neurodegenerative, and even the aging process, are linked to oxidative stress and inflammation. Recently, the Prevention through Mediterranean Diet Study has provided for first time evidence of the benefits of the Mediterranean diet on the primary prevention of cardiovascular disease.

Olive oil, besides its high content of a healthy fat, the monounsaturated (MUFA) one: the oleic acid, has minor components with bioactive properties. The minor components of virgin olive oil are classified into two types: the unsaponifiable fraction, defined as the fraction extracted with solvents after the saponification of the oil, and the soluble fraction which includes the phenolic compounds. The content of the phenolic compounds (polyphenols) of an olive oil depends of the variety of the olive fruit, the cultivar, the climate, the ripeness of the olive, and the type of processing. Virgin olive oils obtained from the first press of centrifugation of the olives are those with high phenolic content. On November 2011, the European Food Safety Authority released a claim concerning the benefits of the daily ingestion of olive oil rich in phenolic compounds, such as the virgin olive oil. Due to this, the need to optimize the olive oil processing in order to obtain high phenolic content olive oils is one of the current goals in terms of increasing the nutritional value of an olive oil. To obtain an optimized olive oil with high phenolic content (OHPCO) has been one of the achievements within the frame of the NUTRAOLEOUM Project.

However, the healthy properties of the new olive oils (OHPCO and FOO), according to the Evidence Based Medicine must be tested in proper clinical randomized trials. New olive oil products need to be tested in front of the parental ones (i.e. virgin olive oil obtained by common procedures) in order to ensure that their healthy properties are highlighted. This is the purpose of the NUTRAOLEUM Study. In order to be able to obtain future health claims from EFSA or FDA, for the products, the investigators will also examine the bioavailability in humans of the active principles (phenolic compounds and triterpenes) of the olive oils, as well as possible basic mechanisms involved in the potential health benefits of the olive oils tested.

DETAILED DESCRIPTION:
The Mediterranean diet, in which olive oil is the main source of fat, has shown to be protective for chronic degenerative diseases. These diseases, such as cardiovascular, cancer, and neurodegenerative, and even the aging process, are linked to oxidative stress and inflammation. Recently, the Prevention through Mediterranean Diet Study has provided for first time evidence of the benefits of the Mediterranean diet on the primary prevention of cardiovascular disease. In human, randomized, controlled studies olive oil, and particularly the virgin one rich in phenolic compounds, have been shown to provide benefits on oxidative damage, inflammation, and on the generation of cell adhesion molecules, a key process for atherosclerosis development.

Olive oil, besides its high content of a healthy fat, the monounsaturated (MUFA) one: the oleic acid, has minor components with bioactive properties. The minor components of virgin olive oil are classified into two types: the unsaponifiable fraction, defined as the fraction extracted with solvents after the saponification of the oil, and the soluble fraction which includes the phenolic compounds. The content of the phenolic compounds (polyphenols) of an olive oil depends of the variety of the olive fruit, the cultivar, the climate, the ripeness of the olive, and the type of processing. Virgin olive oils obtained from the first press of centrifugation of the olives are those with high phenolic content. On November 2011, the European Food Safety Authority (EFSA, 2011) released a claim concerning the benefits of the daily ingestion of olive oil rich in phenolic compounds, such as the virgin olive oil. The Panel considers that in order to bear the claim, 5 mg of hydroxytyrosol and its derivatives (e.g. oleuropein complex and tyrosol) in olive oil should be consumed daily. These quantities, if provided by moderate amounts of olive oil, can be easily consumed in the context of a balanced diet (EFSA, 2011). The conditions for the use of the claim in the bottles, are regulated in the Commission Regulation (EU).Nº 432/2012 of 16 May 2012 (Official Journal of the European Union , L136/1. 25, 5, 2012). According to this regulation: "The claim may be used only for olive oil which contains at least 5 mg of hydroxytyrosol and its derivatives (e.g. oleuropein complex and tyrosol) per 20 g of olive oil. In order to bear the claim, information shall be given to the consumer that the beneficial effect is obtained with a daily intake of 20 g of olive oil". This implies that only high phenolic content olive oils can bear the claim. Due to this, the need to optimize the olive oil processing in order to obtain high phenolic content olive oils is one of the current goals in terms of increasing the nutritional value of an olive oil. To obtain an optimized olive oil with high phenolic content (OHPCO) has been one of the achievements within the frame of the NUTRAOLEOUM Project. In this sense we must point out that, among minor olive oil components, not only polyphenols, but components of the unsaponifiable fraction such as the triterpenes have also shown to have potential for providing benefits for health. The seeds and the skin of the olives, used to produce pomace olive oil, are very rich in triterpenes. Pomace olive oil and triterpenes, such as oleanolic and maslinic acids, have shown anti-inflammatory, antioxidant, and vasodilatation properties in cellular and animal models. Due to this, the enrichment of an OHPCO with olive triterpenes, by joining the healthy properties of virgin and pomace olive oil, will result in a Functional Olive Oil (FOO) with a high bioactive potential for health. This FOO has also been developed in the frame of the NUTRAOLEUM Project. Consumers are every day asking for an "added value" in the nutritional properties of the food to be purchased and responses from the Olive Oil Industry are needed.

However, the healthy properties of the new olive oils (OHPCO and FOO), according to the Evidence Based Medicine must be tested in proper clinical randomized trials. New olive oil products need to be tested in front of the parental ones (i.e. virgin olive oil obtained by common procedures) in order to ensure that their healthy properties are highlighted. This is the purpose of the NUTRAOLEUM Study. In order to be able to obtain future health claims from EFSA or FDA, for the products, we will also examine the bioavailability in humans of the active principles (phenolic compounds and triterpenes) of the olive oils, as well as possible basic mechanisms involved in the potential health benefits of the olive oils tested.

ELIGIBILITY:
Inclusion Criteria:

* healthy on the basis of physical examination and routine biochemical and hematological laboratory determinations,
* willingness to provide written, informed consent and
* to agree to adherence to the protocol.

Exclusion Criteria:

* smoking,
* intake of antioxidant supplements,
* aspirin, or any other drug with established antioxidant properties,
* hyperlipemia,
* obesity (body mass index >30 kg/m2),
* diabetes,
* hypertension,
* celiac or other intestinal disease,
* any condition limiting mobility,
* life-threatening diseases, or
* any other disease or condition that would impair compliance.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2014-02; Primary Completion 2016-06 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Systolic and diastolic blood pressures | Up to 10 months
  measured with a mercury sphygmomanometer after a minimum of 10 minutes rest in the seated position; the average of two measurements was taken for analysis.
Physical activity | Up to 10 months
  a potential confounder variable concerning oxidative and anti-inflammatory status was recorded at the beginning and at the of the study, and assessed by the Minnesota Leisure Time Physical Activity Questionnaire validated for its use in Spanish men and women
Serum glucose | Up to 10 months
  determined by enzymatic methods
Total cholesterol | Up to 10 months
  determined by enzymatic methods
high-density lipoprotein cholesterol | Up to 10 months
  determined by enzymatic methods
triglycerides | Up to 10 months
  determined by enzymatic methods
LDL cholesterol | Up to 10 months
  calculated by the Friedewald formula
Oxidized LDL (oxLDL) | Up to 10 months
  determined in plasma by ELISA using two antibodies against antigenic determinants of oxidized apolipoprotein B molecule (ox-LDL, Uppsala, Sweden)
Conjugated dienes in LDL | Up to 10 months
  measured spectrophotometrically at 234 nm and 300 nm after Cu++ oxidation
Tyrosol and hydroxytyrosol in urine samples and oleanolic and maslinic in plasma | Up to 10 months
  measured as markers of compliance of the intervention, will be determined by gas chromatography-mass spectrometry

SECONDARY OUTCOMES:
Endothelial Function | Up to 10 months
  Endothelial function was measured at baseline (0h) and at 4 and 6h after each olive oil administration. Peripheral arterial tonometry signals were obtained using a device. Finger probes were placed on the middle finger of each subject's hand. These probes comprised a system of inflatable latex air cuffs connected by pneumatic tubes to an inflating device controlled through a computer algorithm. A constant counter pressure (pre-determined by baseline diastolic blood pressure) was applied. There was no occlusion of arterial blood flow. Pulsatile volume changes of the distal digit induced pressure alterations in the finger cuff, which were sensed by pressure transducers and transmitted to and recorded by the device. A decrease in the arterial blood volume in the distal finger tip caused a decrease in pulsatile arterial column changes, reflected as a decrease in the measured PAT signal.

CONTACTS AND LOCATIONS:
Overall Officials: BLAS GIL, Doctor, Principal Investigator — Medical doctor; Montse Fito, Doctor, Principal Investigator — Head of Research Group; Emilo Martínez, Principal Investigator — Head of Research Group
Locations (1):
- University Hospital Virgen de las Nieves, Granada, Granada, Spain

REFERENCES:
- [Derived] Sanchez-Rodriguez E, Biel-Glesson S, Fernandez-Navarro JR, Calleja MA, Espejo-Calvo JA, Gil-Extremera B, de la Torre R, Fito M, Covas MI, Vilchez P, Alche JD, Martinez de Victoria E, Gil A, Mesa MD. Effects of Virgin Olive Oils Differing in Their Bioactive Compound Contents on Biomarkers of Oxidative Stress and Inflammation in Healthy Adults: A Randomized Double-Blind Controlled Trial. Nutrients. 2019 Mar 6;11(3):561. doi: 10.3390/nu11030561. PMID 30845690
- [Derived] Sanchez-Rodriguez E, Lima-Cabello E, Biel-Glesson S, Fernandez-Navarro JR, Calleja MA, Roca M, Espejo-Calvo JA, Gil-Extremera B, Soria-Florido M, de la Torre R, Fito M, Covas MI, Alche JD, Martinez de Victoria E, Gil A, Mesa MD. Effects of Virgin Olive Oils Differing in Their Bioactive Compound Contents on Metabolic Syndrome and Endothelial Functional Risk Biomarkers in Healthy Adults: A Randomized Double-Blind Controlled Trial. Nutrients. 2018 May 16;10(5):626. doi: 10.3390/nu10050626. PMID 29772657
- [Derived] Biel S, Mesa MD, de la Torre R, Espejo JA, Fernandez-Navarro JR, Fito M, Sanchez-Rodriguez E, Rosa C, Marchal R, Alche JD, Exposito M, Brenes M, Gandul B, Calleja MA, Covas MI. The NUTRAOLEOUM Study, a randomized controlled trial, for achieving nutritional added value for olive oils. BMC Complement Altern Med. 2016 Oct 22;16(1):404. doi: 10.1186/s12906-016-1376-6. PMID 27770787
- See also: Related Info — http://www.fibao.es/